CLINICAL TRIAL: NCT05492487
Title: A Pilot Study on Fertility Conservative Treatment of Atypical Endometrial Hyperplasia in Singapore
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Phoon Wai Leng Jessie, Assistant Professor, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB 2019/2551
Record Dates: First submitted 2022-04-07; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Endometrial Hyperplasia; Fertility Issues; Disease Regression; Treatment Side Effects
Keywords: Endometrial Hyperplasia; Fertility; Disease Regression; Randomised Clinical Trial; Mirena IUS; Megace
MeSH Terms: conditions — Endometrial Hyperplasia; Infertility | interventions — Levonorgestrel; Megestrol Acetate

STUDY DESIGN:
Intervention Model Description: Participants will be randomised into either the megace group or the Mirena group. There will be sealed envelopes containing a paper with either Mirena or megace printed on each of them. Participants can chose an envelope at random. The patient and PI will not be blinded of the selection in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirena Arm (Experimental): The patients in the Mirena arm will have a Mirena inserted at time of recruitment of the study. An endometrial biopsy will be performed to assess for disease progression, regression or persistence after 3 months. The endometrial biopsy will be performed via bedside endometrial sampling or hysteroscopic biopsy. As Mirena can be used for treatment of atypical hyperplasia as well as endometrial protection (decreases the risk of endometrial hyperplasia recurrence), the option of keeping or changing the Mirena during biopsy will be discussed with the patient.
  Interventions: Drug: Mirena
- Megace Arm (Experimental): The patients in the megace arm will have be prescribed 3 months of oral megace at time of recruitment of the study. An endometrial biopsy will be performed to assess for disease progression, regression or persistence after 3 months. The endometrial biopsy will be performed via bedside endometrial sampling or hysteroscopic biopsy.
  Interventions: Drug: Megace

INTERVENTIONS:
Drug: Mirena — Mirena Intrauterine System (Mirena-IUS) is a levonorgestrel-releasing intrauterine system. Mirena consists of a T-shaped polyethylene frame (T-body) with a steroid reservoir (hormone elastomer core) around the vertical stem. The reservoir consists of a white or almost white cylinder, made of a mixture of levonorgestrel and silicone (polydimethylsiloxane), containing a total of 52 mg levonorgestrel. Mirena is approved for intrauterine contraception and in 2009 to treat heavy periods for women who choose intrauterine contraception. Mirena is often used off-label for the treatment of endometrial hyperplasia. Levonorgestrel is a progestogen used in a variety of contraceptive products. Low doses of levonorgestrel can be administered into the uterine cavity with the Mirena intrauterine delivery system. Mirena has mainly local progestogenic effects in the uterine cavity.
  Arms: Mirena Arm
Drug: Megace — Megestrol acetate (Megace) is a synthetic derivative of the natural occurring steroid hormone, progesterone. It is licensed for the treatment of anorexia, cachexia or unexplained weight loss in patients with a diagnosis of acquired immunodeficiency syndrome (AIDS) and palliative treatment of advanced breast or endometrial cancer. Megace is often used off-label for the treatment of endometrial hyperplasia. While the precise mechanism by which Megace produces its antineoplastic effects against endometrial carcinoma and endometrial hyperplasia is unknown at the present time, inhibition of pituitary gonadotrophin production and resultant decrease in estrogen secretion may be factors. There is evidence to suggest a local effect as a result of the marked changes brought about by the direct instillation of progestational agents into the endometrial cavity.
  Arms: Megace Arm

SUMMARY:
The investigators' objective is to determine the regression rate, side effects and acceptability of Mirena compared to megace in the treatment of atypical endometrial hyperplasia among women desiring fertility.

DETAILED DESCRIPTION:
Atypical endometrial hyperplasia is a growing clinical problem that increases the risk of carcinogenesis and negatively impacts fertility. Although oral medical treatment may lead to regression in up to 90% of patients, they are associated with adverse side effects such as weight gain, that negatively affects fertility. To-date, there has been no RCTs evaluating the performance of the Mirena Intrauterine System (IUS) with megestrol acetate (megace) (the most effective and commonly used progestogen) in treating women with atypical hyperplasia who still desire fertility.

ELIGIBILITY:
Inclusion Criteria:

* All women diagnosed with atypical hyperplasia aged 21 years to 40 years
* Keen for fertility-preserving treatment

Exclusion Criteria:

* Patients who are currently undergoing treatment for atypical hyperplasia
* Patients with a history of endometrial carcinoma

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Regression | Review in 3 months, maximum up to 9 months of treatment.
  Participants will be reviewed in clinic every 3 months. An endometrial biopsy via hysteroscopy or bedside endometrial sampling will be performed to assess persistence, progression or resolution of the disease.
Time taken for regression of the disease | Review in 3 months, maximum up to 9 months of treatment.
  Participants will be reviewed in clinic every 3 months. An endometrial biopsy via hysteroscopy or bedside endometrial sampling will be performed to assess persistence, progression or resolution of the disease.

SECONDARY OUTCOMES:
Patient Acceptability | Review in 3rd months.
  Number of participants who are keen to continue their current treatment or change the treatment, at the end of 3rd months follow-up.
Patient Acceptability | Review in 6th months.
  Number of participants who are keen to continue their current treatment or change the treatment, at the end of 6th months follow-up.
Patient Acceptability | Review in 9th months.
  Number of participants who are keen to continue their current treatment or change the treatment, at the end of 9th months follow-up.
Side Effects | Through study completion, an average of 9 months.
  Number of participants with side effects such as irregular bleeding, nausea/bloatedness or acne.

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goh CSY, Loh MJM, Lim WW, Ang JX, Nadarajah R, Yong TT, Tong P, Yeo YC, Phoon JWL. A multi-centre randomised controlled trial comparing megestrol acetate to levonorgestrel-intrauterine system in fertility sparing treatment of atypical endometrial hyperplasia. J Assist Reprod Genet. 2024 Sep;41(9):2485-2494. doi: 10.1007/s10815-024-03172-z. Epub 2024 Aug 31. PMID 39215793